CLINICAL TRIAL: NCT06669104
Title: Thoracic Surgery by the Medtronic Hugo™ Robotic System: a Prospective Single Centre Study
Brief Title: Thoracic Surgery by the Medtronic Hugo™ Robotic System
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Calvin Sze Hang Ng, Professor, Chinese University of Hong Kong
Other Study IDs: CUHK HUGO
Record Dates: First submitted 2024-10-16; First posted 2024-11-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Thoracic Cancer
Keywords: robotic assisted thoracic surgery; minimally invasive surgery; lung cancer; mediastinal tumour
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lung specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Lobectomy , Segmentectomy Wedge resection of lung
  Interventions: Device: Medtronic Hugo™ surgical robotic system
- Anterior Mediastinal Tumour Resection
  Interventions: Device: Medtronic Hugo™ surgical robotic system
- Posterior Mediastinal Tumour Resection
  Interventions: Device: Medtronic Hugo™ surgical robotic system

INTERVENTIONS:
Device: Medtronic Hugo™ surgical robotic system — undergoing robotic thoracic surgery by the Medtronic Hugo™ surgical robotic system

SUMMARY:
The introduction of robot-assisted surgery is one of the biggest breakthroughs in surgery, and represents the most significant advancement in minimally invasive surgery of recent decades. One of the first surgical uses of the robot was in orthopaedics, neurosurgery and cardiac surgery. However, it's use has now been well recognized in thoracic surgical procedures ranging from mediastinal tumour resection to complex major lung resections.

Robotic surgery by the da Vinci Surgical System (Intuitive Surgical, Inc) has been one of the most commonly used robotic systems in surgery. The robotic system overcomes the limitations of the standard thoracoscopic approach and allows for precise dissection in a confined space. These advantages include stable operator-controlled camera, high- definition 3D magnified view of 10 to 12 times, articulating instruments with seven degrees of freedom, motion scaling, and tremor filtration.

Recently the Medtronic Hugo™ surgical robotic system has passed the CE mark. This robotic platform, made up of modular surgical arms on wheeled carts, has started its operation in human in Latin America, Europe and the Asia-Pacific region. The Hugo™ system is designed to provide a lower barrier to entry for hospitals looking to expand their reach in robotic surgery. Compared to the platform by Intuitive Surgical, Hugo™can be customized with up to four independent arms, and rolled to different locations in a hospital when needed.

The investigator's centre is the first robotic surgical centre in Hong Kong since 2005. Over the years, the investigator have established the centre to be one of the leading centre in Hong Kong and the region, with involvement in various new development in thoracic robotic procedures, publications and books, and more recently in robotic endo-lumenal procedures.

In this study, the investigator evaluate the early surgical outcome and objective functional outcome of patients undergoing robotic thoracic surgery by the Medtronic Hugo™ surgical robotic system.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 - 80 years
2. Body mass index <35 kg/m2
3. Suitable for minimally invasive surgery
4. Willingness to participate as demonstrated by giving informed consent

Exclusion Criteria:

1. Contraindication to general anaesthesia
2. Severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic intervention
3. Untreated active infection
4. Non-correctable coagulopathy
5. Emergency surgery
6. Vulnerable population (e.g. mentally disabled, pregnancy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are advised to have robotic thoracic procedures
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
The conversion rate | 1 year
  The feasibility of the Medtronic Hugo™ robotic system for thoracic robotic procedures (anterior mediastinal tumour resection, posterior mediastinal tumour resection and lung resection (wedge, segmentectomy, lobectomy), as measured by the conversion rate
The peri-operative complication | 1 year
  The safety profile of the Medtronic Hugo™ robotic system for thoracic robotic procedures (anterior mediastinal tumour resection, posterior mediastinal tumour resection and lung resection (wedge, segmentectomy, lobectomy), as measured by the peri-operative complication profile.

SECONDARY OUTCOMES:
Completeness of Resection evaluated by histopathological analysis | 1 month
  Evaluated by assessing whether the surgical margins are free of tumor as determined by histopathological analysis.
  If the tumor is not touching the resection margins, it is considered a complete resection; If tumor cells are present at the margins, this indicates an incomplete resection.
Resection margin measured by histopathological methods | 1 month
  Measured in millimeters by histopathological methods, indicating the distance from the tumor to the closest margin.
Number of Lymph Nodes Harvested assessed through pathological examination | 1 month
  Total count of lymph nodes excised during the procedure, assessed through pathological examination.
Clinical Recurrence investigated through follow-up imaging | 1 year
  Clinical Recurrence: Monitored through follow-up imaging and clinical evaluations at specified time intervals to determine any recurrence of the disease
  Local recurrence rate (for cancer surgery) will be calculated using the Kaplan-Meier method, and differences between groups will be compared using the log-rank test. A 2-sided P value <0.05 is considered to be statistically significant.
Functional outcome (pre and post lung function test) will be collected | 1 year
  The functional outcomes for lung resection procedures (wedge, segmentectomy, lobectomy) will be assessed by conducting lung function tests. The following parameters will be measured:
  Pulmonary Function Tests (PFTs):
  Forced Vital Capacity (FVC): Measures the maximum amount of air a person can forcibly exhale after taking a deep breath, the measure unit is Liter.
  Forced Expiratory Volume in 1 second (FEV1): Measures the amount of air a person can forcibly exhale in one second, the measure unit is Liter.
  Diffusion Capacity for Carbon Monoxide (DLCO): Assesses how well oxygen and carbon dioxide are exchanged in the lungs, the measure unit is ml/min/mm Hg.

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Sze Hang Ng, Principal Investigator — CUHK
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided